CLINICAL TRIAL: NCT04278430
Title: Does Transcranial Direct Current Stimulation Affect Selective Visual Attention in Children With Left-sided Infantile Hemiplegia? A Preliminary Randomized Controlled Study
Brief Title: Transcranial Direct Current Stimulation for Attention Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, faizan kashoo, PT, Prinicipal investigator, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-1441-78
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Infantile Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The care provider were masked and the pre-post testing was performed by different therapist unaware of the assignment of children.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real tDCS group (Experimental): The tDCS applied over dorsolateral prefrontal cortex for 20 minutes with 1.5 mA intensity
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): The tDCS applied over dorsolateral prefrontal cortex for 20 minutes with 0 mA intensity.
  Interventions: Device: Sham tDCS
- Control (Active Comparator): The normal heathy children age matched undergo the same activity and brain stimulation as the real tDCS group.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — The tDCS stimulator (ActivaDose II tDCS Device; IOMED Inc., Salt Lake City, USA) is a standardized instrument used and tested in children. Two tDCS electrodes of dimensions 3" x 3" were used for the brain stimulation. The electrodes were inserted into a wet saline sponge.
  Arms: Control; Real tDCS group
Device: Sham tDCS — Five children with LSIH were randomly allocated to this group. All participants received sham tDCS for 3 weeks on alternate days and completed 10 treatment sessions. The sham tDCS followed preparatory procedures similar to that used for the experimental group, except that the device was disconnected after the initial increase of the current. Children usually started the activity without noticing that the device was disconnected. The children were assessed at baseline, during the 5th and 10th sessions, and during a follow-up that was scheduled for 4 months later.
  Arms: Sham tDCS

SUMMARY:
Infantile hemiplegia due to brain injury is associated with poor attention. Left-sided infantile hemiplegia affects the learning and acquisition of new skills. This study is aiming to improve the Selective visual attention (SVA) through transcranial direct current stimulation (tDCS) in children with Left-sided infantile hemiplegia .

DETAILED DESCRIPTION:
Infantile hemiplegia (IH) refers to brain injuries that occur before or at birth and lead to hemiplegia/ total paralysis of one side of the body, including the face, arm and leg. The IH is quit rare condition and occurs in 1 in 1000 live births. however, the condition is reported to cause functional and cognitive disability. Children with IH suffer from poor attention particularly visual attention, that is essential to be understand the written language. A focused reading is essential in learning and children with IH possess moderate intelligence and attend school.

Transcranial direct current stimulation(tTCS) is a novel intervention that use small amplitude electrical currents to stimulate the essential areas of the brain through surface electrodes placed on the corresponding areas of the brain.

The eligible children were divided into two groups. one group received tDCS with visual attention activities and the second group received sham tDCS with similar activities. The effect will be assessed before and after with Strops-color testing and a academic reading test.

The experiment intends to explore the affect of tTCS on visual attention span among children with Left-sided infantile hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8-15 years
* Left-sided infantile hemiplegia
* lesion to non-dominant hemisphere

Exclusion Criteria:

* History of epilepsy
* second stroke
* color blind
* under medication for psychiatric illness

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
The Computerized Stroop Color-Word Test | 3 weeks
  The Computerized Stroop Color-Word Test consists of two phases.The first phase is the preparation phase, where the children are asked to identify the color of a circle on the monitor (red, blue, green, or yellow) and press the corresponding key on the keyboard using the unaffected side. Scores obtained at this stage were not included in the final results. The second phase is the actual test, which consists of 96 colorful words, divided into 48 correctly matched colorful words and 48 incorrectly matched colorful words. The words that appeared on the computer screen were presented in a randomized sequence. Each word appeared on the computer screen for 2000 ms with an 800-ms interval. The children were asked to identify the color of the words regardless of their meanings.

SECONDARY OUTCOMES:
academic practical test | 3 weeks
  An academic practical test will be needed to evaluate the improvement in SVA among children. Therefore, a reading comprehension test will be added to the outcome variables. All the three groups performed a reading comprehension test at the baseline, during the 5th and 10th sessions, and during the follow-up period. Two different stories (unread before and equal difficulty) will be selected from their English course and presented to them at the start and following the completion of the 10th session. These stories comprised of between 700 and 1000 words and the time allowed to complete the story was 20 minutes. In the end, the children were asked to answer 10 multiple-choice questions (MCQ) related to the story. Each correct answer will be assigned 1 point.

IPD SHARING:
Plan to Share IPD: Undecided
The Data sharing depends on the permission from the parents of the children and research team.